CLINICAL TRIAL: NCT03291249
Title: A Randomized, Placebo-controlled ,Double-blind, Phase IIa Assessment of the Safety of Foralumab, an Oral Anti-CD3 Antibody, in Patients With Nonalcoholic Steatohepatitis (NASH) and Type 2 Diabetes Mellitus (T2DM)
Brief Title: Assessment of the Safety of Foralumab, an Oral Anti-CD3 Antibody, in Patients With NASH and T2DM
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to MOH request.
Sponsor: Tiziana Life Sciences LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TZLS-0401-001
Record Dates: First submitted 2017-08-21; First posted 2017-09-25 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2017-08

CONDITIONS: NASH - Nonalcoholic Steatohepatitis; NAFLD; T2DM (Type 2 Diabetes Mellitus)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2 | interventions — foralumab; Muromonab-CD3; Omeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Placebo Comparator): Group A will receive placebo solution for 30 consecutive days
  Interventions: Other: placebo; Drug: Omeprazole 20mg
- Group B (Experimental): Group B will receive 0.5 mg Foralumab Solution daily for 30 consecutive days
  Interventions: Drug: Foralumab; Drug: Omeprazole 20mg
- Group C (Experimental): Group B will receive 2.5 mg Foralumab Solution daily for 30 consecutive days
  Interventions: Drug: Foralumab; Drug: Omeprazole 20mg
- Group D (Experimental): Group B will receive 5.0 mg Foralumab Solution daily for 30 consecutive days
  Interventions: Drug: Foralumab; Drug: Omeprazole 20mg

INTERVENTIONS:
Drug: Foralumab — Anti CD3 mAb
  Other Names: Anti CD3
  Arms: Group B; Group C; Group D
Other: placebo — Placebo oral solution
  Arms: Group A
Drug: Omeprazole 20mg — Omeprazole is a proton pump inhibitor used to neutralize stomach PH

SUMMARY:
This is a randomized, placebo-controlled, four-arm, double-blind study. Subjects will be randomized (1:1:1:1) to receive either a daily oral placebo solution or a daily oral dose of 0.5 mg, 2.5 mg or 5.0 mg Foralumab Solution for 30 consecutive days. Subjects will record adverse events and daily administration of study medication in a subject diary. This will serve as a measure of compliance and record of safety and tolerability. Subjects will be followed up for 30 days following completion of treatment.

Study visits performed on Days 14, 30 and 60 of the study, will monitor metabolic parameters (body mass index [BMI] and waist circumference), serum lipid profiles, immunological markers (c-reactive protein [CRP] and an array of cytokines), hepatic enzymes and functions (13C-methacetin breath test [MBT]) and liver steatosis/fibrosis, which will be compared to baseline levels (Day 1).

The safety and tolerability of the treatment regimen will be determined by monitoring vital signs, laboratory values, adverse events and physical findings throughout the study. In addition, its efficacy will be established upon either reduced Day 30 serum alanine aminotransferase (ALT) levels, reduced hemoglobin A1c (HbA1c) or improved homeostasis model assessment (HOMA) or HOMA of insulin resistance (HOMA-IR) scores as compared to baseline (Day 1). In addition, to assess the efficacy of the tested Foralumab Solution regimen in improving overall subject status, a battery of exploratory metabolic, immunologic and hepatic markers will be evaluated on Days 30 and 60.

DETAILED DESCRIPTION:
A randomized, placebo-controlled, double-blind, phase IIa study for assessment of the safety of Foralumab, an oral anti-CD3 antibody, in patients with nonalcoholic steatohepatitis (NASH) and type 2 diabetes mellitus (T2DM).

This is a randomized, placebo-controlled, four-arm, double-blind study. Subjects will be randomized (1:1:1:1) to receive either a daily oral placebo solution or a daily oral dose of 0.5 mg, 2.5 mg or 5.0 mg Foralumab Solution for 30 consecutive days. Subjects will record adverse events and daily administration of study medication in a subject diary. This will serve as a measure of compliance and record of safety and tolerability. Subjects will be followed up for 30 days following completion of treatment.

Study visits performed on Days 14, 30 and 60 of the study, will monitor metabolic parameters (body mass index [BMI] and waist circumference), serum lipid profiles, immunological markers (c-reactive protein [CRP] and an array of cytokines), hepatic enzymes and functions (13C-methacetin breath test [MBT]) and liver steatosis/fibrosis, which will be compared to baseline levels (Day 1).

The safety and tolerability of the treatment regimen will be determined by monitoring vital signs, laboratory values, adverse events and physical findings throughout the study. In addition, its efficacy will be established upon either reduced Day 30 serum alanine aminotransferase (ALT) levels, reduced hemoglobin A1c (HbA1c) or improved homeostasis model assessment (HOMA) or HOMA of insulin resistance (HOMA-IR) scores as compared to baseline (Day 1). In addition, to assess the efficacy of the tested Foralumab Solution regimen in improving overall subject status, a battery of exploratory metabolic, immunologic and hepatic markers will be evaluated on Days 30 and 60.

Primary: To assess the safety and tolerability of the tested Foralumab Solution regimen in subjects with both T2DM and NASH/NAFLD Secondary: To assess the efficacy of the tested Foralumab Solution regimen in improving serum ALT levels, HbA1c, HOMA or HOMA-IR scores in subjects with both T2DM and NASH/NAFLD.

Exploratory: To assess the efficacy of the tested Foralumab Solution regimen in improving overall subject status, as measured by a battery of metabolic, immunologic and hepatic markers.

48 adult subjects (≥18 years) with T2DM and who meet the inclusion criteria for NASH or NAFLD 2a Up to 25 Foralumab (TZLS-0401) is a fully human IgG1 monoclonal antibody directed against the CD3-epsilon (or CD3ε) antigen expressed on the surface of a type of white blood cell called T-cells, or T-lymphocytes. The Fc region of the antibody is mutated to reduce the cytokine release syndrome associated with parenteral administration of anti CD3. When administered orally, Foralumab is not absorbed and induces a signal at the level of the gut immune system to promote regulatory T cells systemically.

A once-daily oral dose of Foralumab solution (0.5, 2.5 or 5.0 mg) or placebo solution will be taken in the morning on an empty stomach for 30 consecutive days.

Group A will receive placebo solution for 30 days (n=12) Group B will receive 0.5 mg Foralumab Solution daily for 30 days (n=12) Group C will receive 2.5 mg Foralumab Solution daily for 30 days (n=12) Group D will receive 5.0 mg Foralumab Solution daily for 30 days (n=12)

A single 20 mg omeprazole pill will be concomitantly administered daily.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Provision of written informed consent
* Diagnosis of T2DM
* HbA1c < 9.0 while on standard of care
* Historical histology-based confirmation of NASH within 12 months prior to screening OR

Diagnosis of NAFLD based on all the following:

* Presentation of at least one other parameter of the metabolic syndrome from the following list of three:

  (i) hypertension [≥130/85 mmHg or regularly taking an antihypertensive], (ii) dyslipidemia with high serum triglycerides [≥150 mg/dL or regularly taking medicines to lower high triglyceride levels] or low serum HDL [<50 mg/dL for women and <40 mg/dL for men], (iii) obesity (BMI > 30 kg/m2) or central obesity [waistline measurement ≥ 89 cm for women and ≥ 102 cm for men])
* ALT > 40 IU
* Fat fraction >10% in MRI performed during screening or up to 3 months prior to screening.
* Agree to the use of effective contraceptive measures, as defined in the protocol, if either male or female with child-bearing potential.

Exclusion criteria:

* Subject with cirrhosis per biopsy (fibrosis staging score >= 4) or Fibroscan® >14 kPa within 12 months of screening.
* Presence of vascular liver disease
* Any history or evidence of decompensated liver disease such as recurrent variceal bleeding, refractory ascites or hepatic encephalopathy
* Known history of chronic alcoholic liver disease, chronic hepatitis B or C infection, drug-induced liver injury (DILI), hemochromatosis, Wilson's disease, 1-antitrypsin deficiency, primary biliary cirrhosis or secondary sclerosing cholangitis, autoimmune hepatitis
* Known HIV antibody-positive
* History of liver transplantation
* BMI <25kg/m2
* Clinically significant alcohol use
* Score of ≥ 2 on the CAGE questionnaire, OR
* Any subject with current significant alcohol consumption or a history of significant alcohol consumption for a period of more than 3 consecutive months any time within 1 year prior to screening, as determined by medical history (medical chart review and/or interview). Significant alcohol consumption is defined as: females: >20 g/day; males: >30 g/day, with a standard drink in the US averaging 14 g alcohol.
* Type 1 diabetes
* Bariatric surgery within the last 5 years
* Weight loss or gain of ≥5 kg in the past 6 months or >10% change in bodyweight in the past 12 months
* Inadequate vascular access on physical examination
* Lactating/breastfeeding/pregnant at screening
* On an elemental diet or parenteral nutrition
* Concurrent conditions
* Inflammatory bowel disease
* Unstable angina, myocardial infarction, transient ischemic events, or stroke within 24 weeks of screening
* Ongoing infectious disease, excluding recurrent urinary tract infection treated with long-term antibiotic prophylaxis
* Any type of immune-mediated and/or malignant disease
* Any other concurrent condition which, in the opinion of the investigator, could impact adversely on the participating subject or on the interpretation of the study data
* Concurrent medications including:
* Amiodarone taken within 30 days of Day 1 (MBT contraindication)
* Beta-blockers: must be on a stable dose for at least 30 days prior to Day 1 (MBT contraindication)
* Statins: must be on a stable dose for at least 30 days prior to Day 1 (MBT contraindication)
* The following medications taken every day for more than 1 week over the last three months: S-adenosyl methionine (SAM-e), betaine, milk thistle and probiotic supplements (other than yoghurt) with the exception of vitamin E or gemfibrozil, which are allowed

  ** If >= 400 IU vitamin E on a regular basis or gemfibrozil, at any dose, are used, the dose must be stable for more than 3 months;
* immunomodulatory agents including In the last 4 weeks

  * oral or parenteral antibiotics
  * daily treatment with non-steroidal anti-inflammatory drugs (e.g., aspirin (>100 mg/day), ibuprofen, naproxen, imeloxicam, celecoxib)

In the last 3 months

* systemic steroids
* daily treatment with non-steroidal anti-inflammatory drugs (e.g., aspirin (>100mg/day), ibuprofen, naproxen, meloxicam, celecoxib) over 4 or more weeks in the last 3 months
* variable dose of antilipidemic agents (HMG Co-A reductase inhibitors - "statins"). Subjects on stable dose of statins are eligible if missed no more than one week of dosing over the last 3 months

In the last 12 months

o azathioprine, 6-mercaptopurine, methotrexate, cyclosporin, anti-TNF alpha therapies (infliximab, adalimumab, etanercept) or anti-integrin therapies

* Any of the following laboratory abnormalities:
* Neutrophil count ≤1.0 x 109/L
* Platelets <100 x 109/L
* Hemoglobin <10g/dL
* Albumin <3.5g
* International Normalized Ratio (INR) >1.5
* Total bilirubin >1.5 x upper limit of reference range (unless Gilbert's syndrome or extrahepatic source as denoted by increased indirect bilirubin fraction)
* Either creatinine clearance ≤60mL/minute, calculated by Cockroft Gault, or creatinine >1.5x upper limit of reference range
* Regular use of marijuana or marijuana-related products, or use of cocaine, or street drugs, as determined by medical history (medical chart review and/or interview).
* Subjects with symptoms of significant mental illness, inability to cooperate or communicate with the investigator, who are unlikely to comply with the study requirements, or who are unable to provide informed consent.
* Hypersensitivity to methacetin and/or its metabolites (i.e., paracetamol, acetaminophen)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2018-12-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
severity and duration for all adverse events | 30 days after last dose
  Incidence, severity, and duration for all adverse events (AEs), and abnormal laboratory and physical findings up until 30 days after last dose
Abnormal laboratory findings | 30 days after last dose
  Incidence, severity, and duration for all adverse events (AEs), and abnormal laboratory and physical findings up until 30 days after last dose
Abnormal physical findings | 30 days after last dose
  Incidence, severity, and duration for all adverse events (AEs), and abnormal laboratory and physical findings up until 30 days after last dose

SECONDARY OUTCOMES:
Change ALT levels | Day 30 versus Day 1 serum ALT levels
  Day 30 versus Day 1 serum ALT levels
Change in HbA1c levels | Day 30 versus Day 1
  HbA1c levels
change in HOMA/HOMA-IR scores | Day 30 versus Day 1
  Day 30 versus Day 1 change in HOMA/HOMA-IR scores. Insulin and fasting plasma glucose will be measured to calculate HOMA/HOMA-IR

OTHER OUTCOMES:
Body mass index (BMI) | Day 1 versus day 30 and 60
  Measurment of BMI (kg/m^2) Serum lipid profile: total cholesterol, triglycerides, low density lipoprotein (LDL) and high density lipoprotein (HDL) fractions.
Change in Immunological markers | Day 1 versus day 30 and 60
  C-reactive protein (CRP) b. T cell-associated cytokine levels (IL2, 4, 5, 6, 8,10,12, 13, IFN, TNF, TGF c. Regulatory T cell (Tregs) levels (cells positive for: CD4, CD25, CD8, CD56, CD3, CD62, CD127, NKT, FoxP3, LAP)
Cytokine levels | Day 1 versus day 30 and 60
  Measurement of Cytokine levels Mean serum concentrations of, cytokeratin (CK)-18 fragments, C-peptide, glucagon-like peptide-1 (GLP-1), adiponectin c. 13C-Methacetin breath test (MBT) Hepatic steatosis and fibrosis
waist circumference | Day 1 versus day 30 and 60
  measurement of waist circumference (cm)
Serum lipid profile | Day 1 versus day 30 and 60
  Serum lipid concentration will be measured
Regulatory T cell | Day 1 versus day 30 and 60
  Measurement of Regulatory T cell
Liver enzymes | Day 1 versus day 30 and 60
  Measurement of Liver enzymes
Mean serum concentrations of cytokeratin (CK)-18 fragments | Day 1 versus day 30 and 60
  Measurement of (CK)-18 fragments concentration
Mean serum concentrations of C-peptide | Day 1 versus day 30 and 60
  Measurement of C-peptide concentration
Mean serum concentrations of glucagon-like peptide-1 (GLP-1) | Day 1 versus day 30 and 60
  Measurement of glucagon-like peptide-1 (GLP-1) concentration
Mean serum concentrations of adiponectin | Day 1 versus day 30 and 60
  Measurement of adiponectin concentration